CLINICAL TRIAL: NCT01337440
Title: The Efficacy and Safety of Ursodeoxycholic Acid (UDCA) Added to the Dipeptidyl Peptidase-4 Inhibitor, Sitagliptin in People With Type 2 Diabetes and Chronic Liver Diseases
Brief Title: Efficacy and Safety of Ursodeoxycholic Acid (UDCA) Added to the DPP-4 Inhibitor in People With Type 2 Diabetes and Chronic Liver Diseases
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kanazawa University (Other)
Responsible Party: BANYU TOKYO, Merck & Co., Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KanazawaU-1
Record Dates: First submitted 2010-09-16; First posted 2011-04-18 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2011-04

CONDITIONS: Type 2 Diabetes Mellitus; Chronic Liver Disease
Keywords: Ursodeoxycholic Acid; sitagliptin; bile acids; GLP-1
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ursodeoxycholic Acid; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UDCA pretreatment (Active Comparator): Ursodeoxycholic Acid (UDCA) for 12 weeks, then Sitagliptin add-on therapy for additional 12 weeks.
  UDCA dosage: dosing from 600 mg for initial 4 weeks. Then, if there is no adverse effect, UDCA is escalated to 900 mg, po, tid.
  Interventions: Drug: Sitagliptin
- Sitagliptin pretreatment (Active Comparator): Sitagliptin: 50 mg, po, qd for 12 weeks, then UDCA add-on therapy for additional 12 weeks.
  UDCA dosage: dosing from 600 mg for initial 4 weeks. Then, if there is no adverse effect, UDCA is escalated to 900 mg, po, tid.
  Interventions: Drug: UDCA

INTERVENTIONS:
Drug: UDCA — Sitagliptin: 50 mg, po, qd for 12 weeks, then UDCA add-on therapy for additional 12 weeks.
  UDCA dosage: dosing from 600 mg for initial 4 weeks. Then, if there is no adverse effect, UDCA is escalated to 900 mg, po, tid.
  Other Names: Ursodeoxycholic acid (UDCA) goes by the trade names Urso.
  Arms: Sitagliptin pretreatment
Drug: Sitagliptin — UDCA for 12 weeks, then Sitagliptin add-on therapy for additional 12 weeks.
  UDCA dosage: dosing from 600 mg for initial 4 weeks. Then, if there is no adverse effect, UDCA is escalated to 900 mg, po, tid.
  Other Names: Sitagliptin sold under the trade name Januvia
  Arms: UDCA pretreatment

SUMMARY:
1. Objectives

1. To test whether Ursodeoxycholic Acid (UDCA) increases Glucagon-like peptide-1 (GLP-1) response to nutrients and improves glycemic control in people with type 2 diabetes.
2. To test whether sitagliptin enhances UDCA-induced beneficial effect in GLP-1 levels and glycemic control.
3. To test safety of combination therapy of sitagliptin and UDCA in people with type 2 diabetes.

2. Clinical hypothesis.

1. UDCA increases GLP-1 response to nutrients via provoking bile acids excretion from the liver to the intestine/colon.
2. UDCA improves glycemic control in people with type 2 diabetes.
3. Sitagliptin enhances UDCA-induced response of GLP-1 to nutrients.
4. Sitagliptin has additive beneficial effects with UDCA in glycemic control in people with type 2 diabetes.
5. Combination therapy of sitagliptin and UDCA is safe and well-tolerated in people with type 2 diabetes.
6. The combination therapy may loose weight by unique mechanisms of each agent; GLP-1 inhibits appetite by acting on CNS and gastrointestinal motility, whereas UDCA-enhanced circulating primary bile acids increases energy expenditure through the pathway involving G protein-coupled bile acid receptor 1 (Gpbar1, or M-Bar, TGR-5) and subsequent activation of type 2 iodothyronine deiodinase (D2) in brown adipose and muscle tissues, as reported previously.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes
2. HbA1c >=6.5% during 8 weeks prior to the study
3. Treated with none or single oral hypoglycemic agent(OHA: sulfonyl ureas, biguanides, or thiazolidinediones) over 12 weeks prior to the study

Exclusion Criteria:

1. Non-Type 2 diabetes
2. Medical history and/or complication of diabetic ketoacidosis
3. Medical history and/or complication of severe hypoglycemia
4. Insulin treatment within 16 weeks prior to the study
5. Treatment with alpha-glucosidase inhibitors or sitagliptin within 12 weeks prior to the study
6. Treatment with glucocorticoid
7. Unstable glycemic control
8. Hypersensitivity to or contraindication of sitagliptin and voglibose
9. Aspartate transaminase (AST) or alanine transaminase (ALT) >=2.5 time of institutional upper normal limit
10. Uncontrolled hypertension (systolic blood pressure >160mmHg or diastolic blood pressure >100mmHg)
11. Severe health problems not suitable for the study
12. Pregnant or lactating women
13. Hepatitis B or C

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-04; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
the difference of haemoglobin A1c (HbA1c) and glycoalbumin (GA) | 6 months
  the difference of haemoglobin A1c (HbA1c) and glycoalbumin (GA) treating by Ursodeoxycholic Acid (UDCA)or sitagliptin monotherapy, and combination therapy of both two drugs for 3 monthes.

SECONDARY OUTCOMES:
Change from Baseline in Glucagon-like peptide-1 (GLP-1) response to lipid meal test (fat 55%) | 6 months
Change from Baseline in energy expenditure | 6months
Change from Baseline in fasting plasma glucose level | 6months
change from baseline in autonomic nerve function | 6 months
  This is performed by power-spectrum analyses of heart rate variability

CONTACTS AND LOCATIONS:
Locations (1):
- Internal medicine, Kanazawa university hospital, Kanazawa, Ishikawa-ken, Japan

REFERENCES:
- [Background] Sakurai M, Takamura T, Ota T, Ando H, Akahori H, Kaji K, Sasaki M, Nakanuma Y, Miura K, Kaneko S. Liver steatosis, but not fibrosis, is associated with insulin resistance in nonalcoholic fatty liver disease. J Gastroenterol. 2007 Apr;42(4):312-7. doi: 10.1007/s00535-006-1948-. Epub 2007 Apr 26. PMID 17464461
- [Background] Takamura T, Sakurai M, Nakamura M, Shimizu A, Ota T, Misu H, Takeshita Y, Tsuchiyama N, Kurita S, Ando H, Kaneko S. Factors associated with improvement of fasting plasma glucose level by mealtime dosing of a rapid-acting insulin analog in type 2 diabetes. Diabetes Res Clin Pract. 2007 Mar;75(3):278-84. doi: 10.1016/j.diabres.2006.07.019. Epub 2006 Oct 27. PMID 17069922
- [Background] Tsuchiyama N, Takamura T, Ando H, Sakurai M, Shimizu A, Kato K, Kurita S, Kaneko S. Possible role of alpha-cell insulin resistance in exaggerated glucagon responses to arginine in type 2 diabetes. Diabetes Care. 2007 Oct;30(10):2583-7. doi: 10.2337/dc07-0066. Epub 2007 Jul 20. PMID 17644622
- [Result] Hamaguchi E, Takamura T, Sakurai M, Mizukoshi E, Zen Y, Takeshita Y, Kurita S, Arai K, Yamashita T, Sasaki M, Nakanuma Y, Kaneko S. Histological course of nonalcoholic fatty liver disease in Japanese patients: tight glycemic control, rather than weight reduction, ameliorates liver fibrosis. Diabetes Care. 2010 Feb;33(2):284-6. doi: 10.2337/dc09-0148. Epub 2009 Oct 30. PMID 19880582
- [Result] Watanabe M, Houten SM, Mataki C, Christoffolete MA, Kim BW, Sato H, Messaddeq N, Harney JW, Ezaki O, Kodama T, Schoonjans K, Bianco AC, Auwerx J. Bile acids induce energy expenditure by promoting intracellular thyroid hormone activation. Nature. 2006 Jan 26;439(7075):484-9. doi: 10.1038/nature04330. Epub 2006 Jan 8. PMID 16400329
- [Result] Amori RE, Lau J, Pittas AG. Efficacy and safety of incretin therapy in type 2 diabetes: systematic review and meta-analysis. JAMA. 2007 Jul 11;298(2):194-206. doi: 10.1001/jama.298.2.194. PMID 17622601
- [Result] Thomas C, Gioiello A, Noriega L, Strehle A, Oury J, Rizzo G, Macchiarulo A, Yamamoto H, Mataki C, Pruzanski M, Pellicciari R, Auwerx J, Schoonjans K. TGR5-mediated bile acid sensing controls glucose homeostasis. Cell Metab. 2009 Sep;10(3):167-77. doi: 10.1016/j.cmet.2009.08.001. PMID 19723493
- [Result] Lazaridis KN, Gores GJ, Lindor KD. Ursodeoxycholic acid 'mechanisms of action and clinical use in hepatobiliary disorders'. J Hepatol. 2001 Jul;35(1):134-46. doi: 10.1016/s0168-8278(01)00092-7. PMID 11495032
- [Derived] Shima KR, Ota T, Kato KI, Takeshita Y, Misu H, Kaneko S, Takamura T. Ursodeoxycholic acid potentiates dipeptidyl peptidase-4 inhibitor sitagliptin by enhancing glucagon-like peptide-1 secretion in patients with type 2 diabetes and chronic liver disease: a pilot randomized controlled and add-on study. BMJ Open Diabetes Res Care. 2018 Mar 17;6(1):e000469. doi: 10.1136/bmjdrc-2017-000469. eCollection 2018. PMID 29607050